CLINICAL TRIAL: NCT03589508
Title: Testing A Couple-based Program for Alcohol Risk Reduction in the National Guard
Acronym: GF_CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Epstein, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AA023589; R34AA023589 (NIH)
Record Dates: First submitted 2018-06-08; First posted 2018-07-18 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Alcohol; Harmful Use
Keywords: National Guard; Telehealth; Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Sessions: ABCP_P (Experimental): In-person therapy sessions: 6 Weekly Prevention Session conducted in person (half of participants will attend alone, half of participants will attend with a significant other)
  Interventions: Behavioral: In-person sessions: ABCP_P
- Video conference sessions: ABCP_T (Experimental): Video conference therapy sessions: 6 Weekly Prevention Session conducted using videoconference (half of participants will attend alone, half of participants will attend with a significant other)
  Interventions: Behavioral: Video conference sessions: ABCP_T

INTERVENTIONS:
Behavioral: In-person sessions: ABCP_P — 6 weekly sessions of alcohol prevention conducted in person.
  Arms: In-Person Sessions: ABCP_P
Behavioral: Video conference sessions: ABCP_T — 6 weekly sessions of alcohol prevention conducted by video conference.
  Arms: Video conference sessions: ABCP_T

SUMMARY:
The purpose of this project is to develop and test indicated prevention intervention to harness support and health promoting endeavors to address use of alcohol to cope with reintegration challenges in Massachusetts National Guard (MANG) service members.

DETAILED DESCRIPTION:
Specific Aim 1: To modify the existing, efficacious Alcohol Behavioral Couple Therapy (ABCT) manual into a 6-session prevention protocol, called Alcohol Behavioral Couple Prevention (ABCP) that will be developed for delivery via in-person and telehealth platforms. The goal of the new ABCP is for individuals or family dyads to learn to work together to minimize hazardous drinking in order to effectively address other problems often present among returning service members.

Specific Aim 2: To field test feasibility and preliminary efficacy of a prevention protocol using a successive cohort design. First, an in-person protocol will be tested with 4 National Guard (NG) members and then adapt and test the protocol for 4 NG members via an analog telehealth design. Again, the manual and accompanied materials will be revised.

Specific Aim 3: To conduct a small Randomized Controlled Trial (RCT) to compare 2 conditions with 22 NG Members in each: (1) In person (ABCP_P; 11 individual, 11 dyad), and (2) Telehealth (ABCP_T; 11 individual, 11 dyad).

ELIGIBILITY:
Inclusion Criteria for NG member:

* Age 18 and older and a member of the MANG.
* Have a SO or trusted friend who is 18 or older
* Service member endorsed one item on the 10-item Alcohol Use Disorders Identification Test within their lifetime

Exclusion Criteria:

* unable to give consent
* Prisoners
* Principal Investigators determined the participant requires a higher level of care (based on unstabilized psychiatric disorder, and/or high drinking or drug use severity, and/or inability to attend to adl's and/or agitated behavior
* Service Member is unable to read or comprehend English at the 7th grade education level

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Percent Drinking Days | Change from baseline at 2 months post session 1
  Derived from Timeline Followback (TLFB)
Percent Heavy Drinking Days | Change from baseline at 2 months post session 1
  Derived from Timeline Followback (TLFB)
Mean Drinks Per Drinking Day | Change from baseline at 2 months post session 1
  Derived from Timeline Followback (TLFB)
Attitude Items | Baseline and through study completion, about 8 weeks
  6 item self-report questionnaire assessing attitudes toward drinking under different circumstances. Item scores were summed to calculate total scores, with scores ranging from 6 to 24. Higher scores indicate greater attitudes about acceptability of drinking across situations.

SECONDARY OUTCOMES:
Alcohol Expectancies Questionnaire 3 | Change from baseline at 2 months post Session 1
  40 item self-report questionnaire assessing thoughts, feelings and beliefs about alcohol. Sub scale scores are calculated by averaging item scores. Positive expectancy subscales are Global positive, Social and physical pleasure, Social expressiveness, Sexual enhancement, Power and aggression, and Tension reduction and relaxation. Negative expectancy sub scales are Cognitive and physical impairment, and Careless unconcern. Higher scores indicate greater expectancies.
Coping Strategies Scale | Change from baseline at 2 months post Session 1
  25-item brief measure assessing coping in alcohol-specific and non-alcohol situations. Scores range from 1-4 and higher scores indicate greater use of coping skills. Total score is calculated by averaging all values.
World Health Organization Quality of Life (WHOQOL) Questionnaire - Bref | Change from baseline at 2 months post Session 1
  26-item self report assessing quality of life across 4 domains/subscales: Physical health, Psychological, Social relationships, Environment. The first two items measure quality of life and overall health and are examined separately, with scores ranging from 1-5. The four domain scores are calculated by averaging values and scores range from 1-5. Higher scores indicate higher quality of life within each domain. Mean scores are then multiplied by 4 in order to make domain scores comparable with the scores used in the WHOQOL-100 (full scale measure).
Treatment Services Review | Weekly for up to 8 weeks
  Interview assessing quantity and type of services received (e.g., health, psychological) outside of study intervention. Total scores are calculated by summing the number of outside services used. Total scores have a minimum of 0 and no maximum value.
Couple Satisfaction Inventory 16 | Baseline and through study completion, about 8 weeks
  16 item measure assessing satisfaction in couple relationship. Scores range from 0 to 81 and higher scores indicate higher levels of relationship satisfaction. Total score is calculated by summing all values.
Perceived Social Support - Family | Baseline and through study completion, about 8 weeks
  20 item self report assessing perceived level of social support from family members. Higher scores indicate higher level of perceived social support.
Working Alliance Inventory Short Form | Baseline and through study completion, about 8 weeks
  12-item self-report measure of the therapeutic alliance. Total scales are calculated by summing all values. Values range from 1-7 with total scores ranging from 12 to 84). Higher scores indicate greater alliance.
Use of Prevention Skills | Baseline and through study completion, about 8 weeks
  Self-report questionnaire assessing use of skills learned during prevention. Item scores range from 1-5 and a total score is calculated by summing all values. Higher scores indicate greater use of skills.
Outcomes Questionnaire (OQ) - 30 | Baseline and through study completion, about 8 weeks
  30 item self-report questionnaire assessing past week psychological well-being. Scores are summed across items and range from 0 to 120, with higher scores indicating worse psychological well-being.
Copello Coping Questionnaire | Baseline and through study completion, about 8 weeks
  30 item self-report assessing partner alcohol-related coping skill use. Total score is calculated by summing the values from each item and scores range from 0-90 with higher scored indicating greater use of coping strategies.

OTHER OUTCOMES:
Intimate Partner Violence (IPV) | Change from baseline at 2 months post Session 1
  Percent of sample with IPV as determined by scores on the Conflict Screener Form H.
Medical History Questionnaire | Change from baseline at 2 months post Session 1
  40 item self-report assessing presence of medical conditions currently and in the past. Scores are calculated by summing individual item scores with possible scores ranging from 0 to 40. Higher scores indicate greater number of medical problems.
Traumatic Brain Injury (TBI) | Baseline
  Percent of sample with a TBI as determined by scores on the TBI Checklist.
Traumatic Brain Injury (TBI) Checklist | Change from baseline at 4 months post Session 1
  Severity of TBI as determined by total scores on the TBI Checklist. Scores are calculated by summing individual item scores with possible scores ranging from 8 to 88.
End of Prevention Questionnaire | 2 months post Session 1
  Self-report questionnaire of helpfulness of therapy elements on a 7 point scale of -3 (greatly harmful), -2, -1, 0 (neutral), +1, +2, +3 (greatly helpful). Total scores are calculated by averaging scores across individual items.
Client Satisfaction Questionnaire | 2 months post Session 1
  8 item self-report assessing satisfaction with treatment. Individual item scores are averaged to calculate a total score with possible scores ranging from 0 to 4. Two additional items assessed the client's ideal number of sessions and length of treatment, with scores ranging from 1 to 24 sessions and 1-12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Epstein, PhD, Principal Investigator — UMass Worcester
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with researchers outside of the core study team.